CLINICAL TRIAL: NCT04617704
Title: Exploratory Study to Evaluate Efficacy and Safety of GC012F Injection in Chromosomal Abnomalities High-risk BCMA+ Multiple Myeloma
Brief Title: BCMA and CD19 Targeted Fast Dual CART for Chromosomal Abnomalities High-risk BCMA+ Multiple Myeloma
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Changzheng Hospital (Other)
Collaborators: Gracell Biotechnologies (Shanghai) Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Weijun Fu, Director of Hematology Department, Shanghai Changzheng Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GBF003
Record Dates: First submitted 2020-08-20; First posted 2020-11-05 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2020-10

CONDITIONS: Multiple Myeloma
Keywords: high-risk; Fast; Chimeric Antigen Receptor T; BCMA; CD19; Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma; Fasting

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental:GC012F treatment (Experimental): BCMA+ cytogenetic high-risk multiple myeloma patients be treated with a single dose of GC012F cells. Total dose of (1-5)*10^5/kg cells will be administered at Day 0
  Interventions: Biological: GC012F injection

INTERVENTIONS:
Biological: GC012F injection — GC012F injection is a autologous dual CAR-T targeted BCMA and CD19. A single infusion of CAR-T cells will be administered intravenously.

SUMMARY:
This is a single arm, open label, multi-center prospective study to explory the safety and efficacy of GC012F CAR-T cells in patient diagnosed with high-risk chromosomal abnormalities BCMA+ multiple myeloma(MM).

DETAILED DESCRIPTION:
The main aim of this study is to determin the safety and efficacy of GC012F in cytogenetic high-risk MM. GC012F is an autologus dual chimeric antigen receptor T-cell(CAR-T) therapy that targets B-cell maturation antigen(BCMA) and CD19. This study comprises of a screening phase(less than or equal to 28 days prior to apheresis) followed by apheresis(will occur upon enroiiment); Treatment Phase including autologus stem cell transplant on Day-1 followed by infusion of GC012F on Day0 and then post-infusion assessments from Day1 to Day 84; and a Post-treatment Phase(Day 85 and up to end of the study). Efficacy will be explored to assessed and safety will be closely monitored during the study.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of active MM as defined by any of following: a) serum M protein more than or equal to 10g/dL; b) urine M protein more than or equal to 200mg/24 h; c) involved serum free light chain more than or equal to 100mg/dL with abnormal serum kappa lambda ratio;
2. Patients with clear BCMA expression(percent of BCMA positive plasma cells more than or equal to 20%) detected by flow cytometry;
3. High-risk chromosomal abnormal defined as presence of del17p, and/or t(4;14) and/or t(14;16);
4. Estimated life expectancy more than or equal to 3 months;
5. Absolute neutrophil count more than or equal to 1*10^9/L;
6. Platelet count more than or equal to 25*10^9/L;
7. Absolute lymphocyte count more than or equal to 1*10^8/L;
8. Liver, kidney and cardiopulmonary functions meet the following requirements: a) Total bilirubin less than or equal to 2*ULN(except for Gilbert Syndrome); ALT and AST less than or equal to 2.5*ULN, maintenance of kidney function not depend on dialysis; c)Corrected serum calcium less than or equal to 12.5 mg/dL or free ion calcium less than or equal to 6.5mg/dL(1.6mmol/L);
9. Sufficient venous access for leukapheresis collection and no other contraindications to leukapheresis;
10. Subjects and sexual partner with fertility are willing to use effective and reliable method of contraception for at least 1 year after CAR-T infusion;
11. subjects must have signed writtern informed consent.

Exclusion Criteria:

1. Accompanied by other unctrolled maligancies. Two exceptions to this criteria: Recepted radical therapy carcinoma without activity within 3 years before screening; fully treated skin non-melanoma;
2. Any situations not benefit for subjects to accept or tolerated to planned therapy or understand informed consent; or any situation in which investigators believe that participation in this study is not in the subject's best intreat(eg., harm to health), or any situation that may prevent, limit or confuse the assessment;
3. Convulsion or stoke within past 6 months;
4. Any instability or systemic disease within 6 months prior to screening, including but not limited to congestive heart failure(New York heart association classification ≥ III)， unstable angina, cerebrovascular accident, or transient cerebral ischemic, myocardial infarction, LEVF<50%(assessed by an echocardiogram or multi-door circuit scan);
5. Patients have central nervous system(CNS) metastases or CNS involvement(including cranial neuropathies or mass lesions and leptomeningeal disease);
6. Subjects with positive HBsAg or HBcAb positive and peripheal blood HBV-DNA titer is higher than the lower limit of detection of the research institution; HCV antibody positive; HIV antibody positive; syphilis primary screening antibody positive;
7. Presence or suspicious of fungi, bacteria, viruses or other infections that are uncontrollable or requiring intravenous treatment;
8. Activity of autoimmune disease (such as crohn's disease, rheumatoid arthritis, systemic lupus erythematosus), orhistory of autoimmune disease within the last 3 years;
9. Clinical evidence of dementia or changes of mental state;
10. Exist of pulmonary fibrosis;
11. Allergy subjects or history of severe hypersensitivity;
12. Oxgen inhalation requirement to maintain adequate oxygen saturation;
13. Surgery (except for local anesthesia surgery) plan 2 weeks before apheresis, during or 2 weeks after CAR-T infusion;
14. Patients who are accounted to be not appropriate for this investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events after GC012F injection | Minimum 2 years after GC012F infusion

SECONDARY OUTCOMES:
Percentage of MRD negative patients after GC012F infusion | Minimum 2 years after GC012F infusion
ORR(PR, VGPR, CR and sCR) of patients after GC012F treatment | Minimum 2 years after GC012F infusion(Day0)
  percent of subjects who achieving PR or better after GC012F infusion
Progression free survival after GC012F treatment | Minimum 2 years after GC012F infusion(Day0)
Duration of response of subjects after GC012F treatment | Minimum 2 years after GC012F infusion(Day0)
Overall survivalof subjects after GC012F treatment | Minimum 2 years after GC012F infusion(Day0)
Cytokines in serum after GC012F infusion | Minimum 24 weeks after GC012F infusion(Day0)
Subset of lymphocytes in blood after GC012F infusion | Minimum 2 years after GC012F infusion(Day0)
Anti-GC012F antibodies in blood after GC012F infusion | Minimum 2 years after GC012F infusion(Day0)
Cell counts of GC012F in blood and bone marrow(if available) after GC012F infusion | Minimum 2 years after GC012F infusion(Day0)
Copies of GC012F in blood and bone marrow(if available) after GC012F infusion | Minimum 2 years after GC012F infusion(Day0)

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided